CLINICAL TRIAL: NCT05240859
Title: A Multicenter, Prospective, Observational Real World Study For the Efficacy and Safety of a Adalimumab Biosimilar (Geleli) in Rheumatoid Arthritis.
Brief Title: Real World Study of a Adalimumab Biosimilar (Geleli) in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-Z-04
Record Dates: First submitted 2022-02-06; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geleli: RA patients treated with Geleli
  Interventions: Drug: Geleli

INTERVENTIONS:
Drug: Geleli — Adalimumab Biosimilar

SUMMARY:
The purpose of this multicenter, prospective, Observational study is to assess the Efficacy and Safety of an Adalimumab Biosimilar (Geleli) in Rheumatoid Arthritis in the real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants who fulfilled the 1987 revised American College of Rheumatology (ACR) or 2010 ACR/EULAR classification criteria for RA.
* Participants for whom the rheumatologists have decided to initiate Geleli treatment.
* Participants who provide a written informed consent form of participating in this study.

Exclusion Criteria:

* Current active or chronic infections, or previous history of active TB infection.
* History of malignancy.
* Congestive heart failure with NYHA class III or IV.
* Females of childbearing or breastfeeding.
* Participate in other clinical trial within 3 months.
* Allergic to the drugs involved in the study.
* The investigator believes that the patient is not suitable to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RA patients who start Geleli treatment
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving American College of Rheumatology (ACR) 20 | Week 24
  The ACR20 was achieved if there was at least a 20% improvement from baseline in swollen joint count 66 (SJC66) and tender joint count 68 (TJC68) and 3 or more of the 5 following assessments: participant's assessment of pain, GH, physician's global assessment of disease activity, participant's assessment of physical function and CRP.

SECONDARY OUTCOMES:
Percentage of Participants Who Were on Geleli for a Period of 24 Weeks | Week 24
Remission rate According to Boolean Criteria | Week 12 and Week 24
Remission rate According to Clinical Disease Activity Index (CDAI) | Week 12 and Week 24
Proportion of Participants Achieving American College of Rheumatology (ACR) 20 | Week 4 and Week 12
Proportion of Participants Achieving American College of Rheumatology (ACR) 50 | Week 4, Week 12 and Week 24
Proportion of Participants Achieving American College of Rheumatology (ACR) 70 | Week 4, Week 12 and Week 24
Change From Baseline in Disease Activity Score 28 (DAS28)-ESR | Baseline, Week 4, Week12 and Week 24
Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) | Baseline, Week 4, Week12 and Week 24
Assessment of Safety Based on Adverse Events that Occur During the Study. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD, PhD, Principal Investigator — Department of Rheumatology and Immunology, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China